CLINICAL TRIAL: NCT02158611
Title: Whole Person Care Research Program of the Suicide Cases Consultative Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ju Pan, visiting doctor, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 102081-F
Record Dates: First submitted 2014-02-19; First posted 2014-06-09 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Suicide
Keywords: Individual Counseling service; Group Counseling service
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Other)
  Interventions: Other: Lifestyle counseling

INTERVENTIONS:
Other: Lifestyle counseling

SUMMARY:
This project aims to provide more treatment options to suicide patients to further enhance the holistic medical services in Far Eastern Memorial Hospital. It focuses on high-risk cases, especially those whose suicidal behaviors are triggered by interpersonal/or emotional problems because psychological counseling or interpersonal growth groups of services have been shown to be beneficial to this population.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old, survivors from suicide.

Exclusion Criteria:

* under 20 years old
* prisoner
* suffer from a serious illness
* foreigner/ can't speak Chinese
* the people who can't express themselves
* can not be interviewed in FEMH
* people with severe physical or psychological symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
patient's satisficaction questionaire | six weeks
  A form for patients record their comment of each meeting with psychologist and other group member in a supportive group.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan